CLINICAL TRIAL: NCT06794554
Title: A Phase 2, Multicentre, Open-label, Single Arm Study to Evaluate the Effectiveness and Safety of Rezafungin (as Acetate) in the Treatment of Chronic Pulmonary Aspergillosis (CPA) in Patients With Limited Treatment Options
Brief Title: Rezafungin for Treatment of Chronic Pulmonary Aspergillosis (CPA) in Adults With Limited Treatment Options
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR907-2502
Record Dates: First submitted 2024-11-26; First posted 2025-01-27 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pulmonary Aspergillosis
Keywords: Chronic pulmonary aspergillosis; Rezafungin; Rezzayo
MeSH Terms: interventions — Rezafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Rezafungin for Injection, IV, with a 400 mg loading dose on Day 1 of Week 1, followed by 200 mg once weekly, for a total of 26 doses (6 months).
  Interventions: Drug: Rezafungin Acetate

INTERVENTIONS:
Drug: Rezafungin Acetate — IV with a 400 mg loading dose on Day 1 of Week 1, followed by 200 mg once weekly, for a total of 26 doses (6 months).

SUMMARY:
The goal of this clinical trial is to to evaluate the drug rezafungin in the treatment of Chronic Pulmonary Aspergillosis (CPA) in male and female patients aged 18 years and over with limited treatment options.

The study aims to answer whether 6 months of rezafungin treatment is effective and safe in patients with chronic pulmonary aspergillosis with limited treatment options according to clinical and radiological response as measured by the St George's Respiratory Questionnaire, weight, and CT imaging.

Participants will:

* Be given the drug rezafungin every week for 6 months.
* Visit the clinic once a month for checkups and tests.
* Complete questionnaires on thier health and wellbeing.

DETAILED DESCRIPTION:
Chronic pulmonary aspergillosis (CPA) is a progressive and potentially life-threatening fungal infection of the lungs. It is usually, but not exclusively, caused by Aspergillus fumigatus and affects patients with underlying respiratory disorders with a prevalence of less than 1 per 100,000 in Europe. The disease leads to the destruction of lung tissue typified by the insidious enlargement of cavities and fibrosis which can severely impact quality of life and has a mortality of up to 14% in one year. The only approved class of oral antifungals are the azoles such as voriconazole or itraconazole. Treatment with azoles is for a minimum of six months, however, in practice can be long-term and, in some cases, lifelong.

Azole resistance can often be attributed to the suboptimal treatment response rates in CPA. This is possibly a consequence of accumulations of the Aspergillus fungus that form 'aspergillomas' which harbour high concentrations of the fungus, thus driving the propensity to develop resistance. The resistance to one azole can often be associated with pan-azole resistance resulting in a lack of effective oral treatment options.

In addition to drug resistance, azoles are potentially hepatotoxic, can elicit adrenal suppression and neuropathy. One of the main safety concerns with voriconazole is that it has been linked to skin cancer. If azole therapy is not an option due to intolerance or resistance, patients are left with Intravenous (IV) amphotericin B (which due to toxicity can only be given short-term) or IV echinocandins. Currently licensed IV echinocandins need to be given daily which limits the practicality of longer-term therapy.

This proposed study aims to generate clinical data on the efficacy and safety of rezafungin for treatment of CPA.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Males or females ≥18 years of age
3. Established diagnosis of CPA according to ESCMID/ERS criteria (2016) which includes all the following, which should be present for ≥3 months:

   * one or more clinical symptoms (persistent cough, recurrent haemoptysis, weight loss, malaise, night sweats, fever and dyspnoea)
   * slowly progressive or persistent radiological findings (one or more cavities and surrounding fibrosis, infiltrates, consolidation, with or without fungal ball or progressive pleural thickening) on computed tomography (CT) of the thorax
   * immunological, microbiological or molecular evidence of Aspergillus infection (growth of Aspergillus in respiratory secretions or serum galactomannan index >0.5 or BALF galactomannan index >1), positive Aspergillus IgG, or positive PCR
   * exclusion of active tuberculosis or non-tuberculous mycobacterial pulmonary infection or disorders that will prevent evaluation of outcome over 6 months. Patients on anti-mycobacterial therapy can be enrolled if their mycobacterial infection is stabilised
4. Unable to receive systemic azole antifungal therapy due to any of the following: documented or anticipated resistance, intolerance, contraindication (e.g. due to drug-drug interactions or organ dysfunction), inability to take oral medication, or lack of availability. NOTE: the administration of rezafungin is monotherapy only, and subjects currently on azoles who are able to remain on therapy are not eligible
5. Antifungal treatment is indicated according to the opinion of the investigator due to radiological changes consistent with CPA progression OR high burden of symptoms
6. Female subjects of child-bearing potential <2 years post-menopausal (unless surgically sterile) must agree to and comply with using one barrier method (e.g., female condom with spermicide) plus one other highly effective method of birth control (e.g., oral contraceptive, implant, injectable, indwelling intrauterine device, vasectomized partner), or sexual abstinence (only possible if it corresponds to the subject's usual lifestyle) while participating in this study, and for 30 days after the last dose of study drug. Male subjects must be vasectomized, abstain from heterosexual intercourse, or agree to use barrier contraception (condom with spermicide), and agree not to donate sperm while participating in the study and for 120 days from the last IV dose of study drug, unless the partner is >2 years post-menopausal or otherwise sterile.

   * Definitions: Woman of childbearing potential: fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
   * A postmenopausal state: no menses for 12 months without an alternative medical cause.
   * Abstinence: refraining from heterosexual intercourse (only if it corresponds to the subject's usual lifestyle)
7. Willingness to comply with all aspects and assessments required in this study

Exclusion Criteria:

1. Subjects with invasive aspergillosis, aspergillus nodules, or simple aspergilloma
2. Known or suspected hypersensitivity to rezafungin for Injection or any of its excipients
3. Current participation in another interventional treatment trial with an investigational agent. Participation in another interventional treatment trial is permitted during the follow-up period of the study
4. Recent use of an investigational medicinal product within 28 days or 5 half-lives of the investigational medicinal product, whichever is greater, to prevent overlapping toxicities when this study's investigational product is dosed, or presence of an investigational device at the time of screening. In some cases, use of investigational products may be acceptable in consultation with the Sponsor's Medical Monitor
5. Administration of any other echinocandin or intravenous antifungal treatment within 3 months of screening
6. Administration of ≥15mg prednisolone daily (or other equivalent immunosuppressant) for at least 3 weeks within 4 weeks of screening
7. Acute respiratory infections considered inadequately treated in the opinion of the Principal Investigator. Any subjects diagnosed with an acute respiratory infection during the screening period should be re-screened following the required course of appropriate treatment and enrolled when considered adequately treated.
8. Subjects with active malignancy who are receiving chemotherapy or radiation therapy
9. Severely immunocompromising conditions according to the opinion of the investigator such as bone marrow transplantation, neutropenia, or have received cancer chemotherapy within last 6 months
10. Subjects on the palliative care pathway
11. Any other condition or laboratory abnormality that, in the opinion of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with the assessments included in the study
12. A. Meets National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, criteria for ataxia, tremor, motor neuropathy, or sensory neuropathy of Grade 2 or higher B. History of severe ataxia, tremor, or neuropathy or a diagnosis of multiple sclerosis or a movement disorder (including Parkinson's Disease or Huntington's Disease)
13. Planned or ongoing therapy at Screening with a known severe neurotoxic medication or with a known moderate neurotoxic medication in a patient with ataxia, tremor, motor neuropathy, or sensory neuropathy of CTCAE version 5.0 Grade 1 or higher.
14. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in clinical and radiological response at 6 months | 6 months
  Participants achieving a clinical improvement and radioligical improvement by CT scans

CONTACTS AND LOCATIONS:
Locations (37):
- Kepler University Hospital, Linz, Austria
- Belgium (4):
  - Brussels University Hospital, Brussels
  - UZ Gent, Ghent
  - University Hospital Leuven, Leuven
  - CHU UCL Namur, Yvoir
- France (5):
  - CHU Amiens Picardie, Amiens
  - Institut Coeur Poumon CHU, Lille
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Bordeaux, Pessac
  - CHU de Rouen, Rouen
- Germany (3):
  - Evangelische Lungenklinik Berlin, Berlin
  - University of Cologne, Cologne
  - Asklepios Lungenfachklinik Gauting, Gauting
- Országos Korányi Pulmonológiai Intézet, Budapest, Hungary
- Italy (4):
  - University of Genova, San Martino Hospital, Genova
  - University of Pisa, Pisa
  - INMI Lazzaro Spallanzaniconsu, Roma
  - Humanitas Research Hospital, Rozzano
- Radboud Universitair Medisch Centrum Stichting, Nijmegen, Netherlands
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Vall d'Hebron Barcelona Hospital Campus, Barcelona
  - Ramón y Cajal Hospital, Madrid
  - Hospital Sant Joan de Deu de Martorell, Martorell
  - Hospital La Fe, Valencia
- United Kingdom (8):
  - Royal Papworth Hospital, Cambridge
  - University Hospitals of Derby and Burton, Derby
  - Western General Hospital, Edinburgh
  - Leeds Teaching Hospital, Leeds
  - Imperial College Hospital, London
  - Royal Brompton Hospital, Guy's and St. Thomas' Hospital, London
  - University College London (UCL) Hospitals, London
  - Manchester University Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided